CLINICAL TRIAL: NCT02006667
Title: An Open-label Pilot Study Evaluating the Effect of a Combination Regimen of Herceptin, Cisplatin, and Gemcitabine on Time to Disease Progression in Patients With Metastatic Urothelial Cancer
Brief Title: A Study of Herceptin (Trastuzumab) Combination Therapy in Patients With Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17600
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Urinary Tract Cancer
MeSH Terms: conditions — Urologic Neoplasms | interventions — Trastuzumab; Gemcitabine; Cisplatin

ARMS (1):
- Trastuzumab, Gemcitabine, Cisplatin (Experimental): Participants received an initial loading dose of 4 milligrams per kilogram (mg/kg) trastuzumab intravenous (i.v.) on Day 3 of Cycle 1, followed by weekly doses of 2 mg/kg i.v until disease progression; 1200 mg per square meter (m2) gemcitabine i.v. on Days 1, 8, and 15 of Cycles 1 through 6; and 70 mg/m2 cisplatin i.v. on Day 2 of Cycles 1 through 6.
  Interventions: Drug: trastuzumab; Drug: gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: trastuzumab — 4 mg/kg i.v., Day 3 of Cycle 1, followed by weekly doses of 2 mg/kg i.v., Day 1 of Cycle 2 until disease progression
  Other Names: Herceptin
Drug: gemcitabine — 1200 mg/m2 i.v. on Days 1, 8, and 15 of Cycle 1 through 6
Drug: cisplatin — 70 mg/m2 i.v. on Day 2 of Cycles 1 through 6

SUMMARY:
This study will evaluate the efficacy and safety of a chemotherapy regimen of intravenous Herceptin, cisplatin and gemcitabine in patients with metastatic urothelial cancer. The anticipated time on study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with >=18 years of age;
* metastatic urothelial carcinoma;
* measurable metastases or local recurrent disease;
* no prior chemotherapy for metastatic disease;
* HER2 overexpression (IHC [2+] or [3+]).

Exclusion Criteria:

* concomitant chemotherapy or immunotherapy;
* active or uncontrolled infection;
* solely CNS metastases;
* clinically significant cardiac disease, advanced pulmonary disease or severe dyspnoea;
* co-existing malignancies diagnosed within last 5 years, except basal cell cancer or cervical cancer in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2001-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Germany (6):
  - Aschersleben
  - Dessau
  - Fulda
  - Leipzig
  - Marburg
  - Weiden

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab/Gemcitabine/Cisplatin: Participants received gemcitabine 1200 milligrams per square meter (mg/m^2), intravenously (IV), on Days 1, 8, and 15 (for a maximum of six 4-week cycles); cisplatin 70 mg/m^2, IV, on Day 2 (for a maximum of six 4-week cycles); and trastuzumab 4 mg per kilogram (mg/kg), IV, on Day 3 of Cycle 1, followed by weekly doses of 2 mg/kg, IV, until disease progression.
Period: Overall Study
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Started | 13
Completed | 7
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all enrolled participants who received study treatment.
Groups:
- Trastuzumab/Gemcitabine/Cisplatin: Participants received gemcitabine 1200 mg/m^2, IV, on Days 1, 8, and 15 (for a maximum of six 4-week cycles); cisplatin 70 mg/m^2, IV, on Day 2 (for a maximum of six 4-week cycles); and trastuzumab 4 mg/kg, IV, on Day 3 of Cycle 1, followed by weekly doses of 2 mg/kg, IV, until disease progression.
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS was defined as the time from the first dose of study treatment to the first documentation of objective tumor progression or death due to any cause.
Time Frame: Screening, Day 1 of Cycles 1 through 6, every 4 weeks until end of treatment, up to 33 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Number analyzed (Participants) | 13
percentage of participants | 92.3

2. Primary Outcome: Progression-Free Survival - Time to Event
Description: The median time, in months, from the first dose of study treatment to PFS event.
Time Frame: Screening, Day 1 of Cycles 1 through 6, every 4 weeks until end of treatment, up to 33 months
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Number analyzed (Participants) | 13
months | 11.0 [5.7 to 14.3]

3. Primary Outcome: Percentage of Participants Who Were Progression Free at 12 and 24 Months
Time Frame: Screening, and Months 12 and 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Number analyzed (Participants) | 13
percentage of participants
  12 Months | 38.5 [14.1 to 62.8]
  24 Months | 15.4 [2.5 to 38.8]

4. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the start of study treatment to date of death due to any cause.
Time Frame: Screening, Day 1 of Cycles 1 through 6, every 4 weeks until end of treatment, up to 36 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Number analyzed (Participants) | 13
percentage of participants | 84.6

5. Secondary Outcome: Overall Survival - Time to Event
Description: The median time, in months, from the start of study treatment to OS event.
Time Frame: Screening, Day 1 of Cycles 1 through 6, every 4 weeks until end of treatment, up to 36 months
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Number analyzed (Participants) | 13
months | 14.9 [12.9 to 21.7]

6. Secondary Outcome: Percentage of Participants Surviving at 12 and 24 Months
Time Frame: Screening, and Months 12 and 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Number analyzed (Participants) | 13
percentage of participants
  12 Months | 76.9 [44.2 to 91.9]
  24 Months | 23.1 [5.6 to 47.5]

7. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR), Partial Response (PR), or Stable Disease (SD)
Description: Per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1): CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal [(short axis less than (<) 10 millimeters (mm)]. No new lesions. PR was defined as greater than or equal to (≥) 30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. SD was defined as not qualifying for CR, PR, or Progressive Disease (PD).
Time Frame: Screening, Day 1 of Cycles 1 through 6, every 4 weeks until end of treatment, up to 33 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Number analyzed (Participants) | 13
percentage of participants
  CR | 15.4
  PR | 23.1
  SD | 46.2
  PD | 15.4
  CR/PR | 38.5
  CR/PR/SD | 84.6

ADVERSE EVENTS:
Time Frame: Adverse events were reported from randomization until 30 days after the end of treatment.
Description: This study did not include a separate analysis of non-serious AE's. In addition, only events by system organ class were provided, no preferred terms for individual events were available.
Arm/Group | Trastuzumab/Gemcitabine/Cisplatin
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab/Gemcitabine/Cisplatin (N=13)
Tachyarrhythmia (Cardiac disorders) | 1
Gastrointestinal hermorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Chill (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
General disorders-other (General disorders) | 1
Catheter related infection (Infections and infestations) | 1
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab/Gemcitabine/Cisplatin (N=13)
Anemia (Blood and lymphatic system disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Endocrine disorders-other (Endocrine disorders) | 1
Eyelid function disorder (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Chills (General disorders) | 3
Fatigue (General disorders) | 3
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
General disorders and administration site conditions-other (General disorders) | 1
Bronchial infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Infections and infestations-others (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Creatinine increased (Investigations) | 2
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 3
Platelet count decreased (Investigations) | 6
Investigations-other (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified-others (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures-others (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.